CLINICAL TRIAL: NCT00829816
Title: A Multi-Center Phase 1 Study of the Safety and Tolerability of Dimebon in Alzheimer's Disease Patients on Memantine (Cohort 1) and Memantine Plus Donepezil (Cohort 2)
Brief Title: Safety and Tolerability of Dimebon in Patients on Memantine, and Memantine Plus Donepezil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIM17
Record Dates: First submitted 2009-01-12; First posted 2009-01-27 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimers disease; donepezil; memantine
MeSH Terms: conditions — Alzheimer Disease | interventions — latrepirdine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dimebon (Experimental): 20 mg dimebon by mouth 3 times per day
  Interventions: Drug: Dimebon
- Placebo (Placebo Comparator): 20 mg placebo by mouth 3 times per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dimebon
  Arms: Dimebon
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of dimebon given to Alzheimer's disease patients currently on a stable dose and regimen of memantine or memantine plus donepezil.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's disease
* On Memantine
* Caregiver who is willing to accompany the patient to all clinic visits

Exclusion Criteria:

* Unstable medical illnesses or significant hepatic or renal disease
* Other primary psychiatric or neurological disorders

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-12; Primary Completion 2009-04 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of orally administered dimebon in patients with Alzheimer's disease (AD) on a stable dose and regimen of memantine, or memantine plus donepezil. | up to 28 days
  Treatment discontinuation due to adverse events, the frequency and severity of adverse events, and clinically significant changes in safety assessments (including physical examination findings, vital signs, laboratory values, and ECGs) in the dimebon group will be compared to those reported in the placebo group.

SECONDARY OUTCOMES:
To assess the steady-state pharmacokinetics (PK) of orally-administered dimebon in patients with AD on a stable dose and regimen of memantine, or memantine plus donepezil. | up to 28 days
  The following key parameters will be used to assess the steady-state PK of dimebon: maximum plasma concentration (Cmax), time to maximum plasma concentration (tmax), Ctrough, area under the curve (AUC), and peak-to-trough ratio.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Los Alamitos, California
  - National City, California
  - Delray Beach, Florida
  - Orlando, Florida